CLINICAL TRIAL: NCT00344864
Title: A Prospective Clinical Research Project Evaluating The Effects of Soft Contact Lenses on Higher Order Visual Aberrations
Status: Terminated | Type: Observational
Why Stopped: Terminated due to lack of patient recruitment
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Paul Sanchez, MD, UTSW Medical Center at Dallas
Other Study IDs: Sanchez001
Record Dates: First submitted 2006-06-23; First posted 2006-06-27 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2007-05

CONDITIONS: Ocular Refractive Aberrations
Keywords: Contact Lenses Higher Order Aberrations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: LADARWave

SUMMARY:
High order aberrations (HOA) are visual phenomena that decrease quality of vision. Examples of high order aberration are glare, halos, decreased contrast sensitivity and shape distortion. They are caused by slight imperfections or distortions in the corneal surface. HOA are currently measured using a variety of FDA approved devices. For this study, the LADARWave (Alcon) will be used to measure HOA. This device uses a harmless beam of light. It is FDA approved and non-invasive. Contact lens induced high order aberrations have never been measured and reported in the literature. This work may provide information to guide future contact lens design.

DETAILED DESCRIPTION:
Patients will be recruited from the Aston optometry clinic. The pool of patients included in the study will be from those who have voluntarily scheduled appointments for contact lenses. During the patient's initial visit, the study will be explained to them and they will have a choice of whether or not to take part with no penalty for refusal. If a patient agrees to take part in the study, they will have their HOA measured with the LADARWave instrument prior to contact lens insertion and right after contact lens insertion. Patients will then return for visits both one week and one month later for follow up measurements at the time of their regularly scheduled visits.

ELIGIBILITY:
Inclusion Criteria:

All patients of any race and sex between the ages of 18-35 years of age who are not currently wearing contact lenses at their initial presentation. Only patients who voluntarily agree to participate in the study will be included. These potential subjects would be selected after reviewing and signing the Informed Consent (IC) as well as HIPAA authorization forms. The Principal Investigator (PI) or his designee will introduce the study to the patient, thoroughly explaining the details of the study. Copies of the forms will be placed in the patient medical record as well as given to study patient.

Exclusion Criteria:

Patients under the age of 18 or over the age of 35 will be excluded. Patients with any ocular pathology, previous eye surgery and/or uveitis will be excluded. Also, any patient who does not choose to participate will be excluded.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All patients of any race and sex between the ages of 18-35 years of age who are not currently wearing contact lenses at their initial presentation.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2006-01; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Whether Soft contact lenses induce High order aberrations (HOA)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sanchez, MD, Principal Investigator — UTSW Medical Center At Dallas; James McCulley, MD, Study Chair — UTSW Medical Center Dallas
Locations (2):
- United States (2):
  - Aston Ambulatory Care Center, Dallas, Texas
  - UTSW Medical Center At Dallas, Dallas, Texas